CLINICAL TRIAL: NCT02445040
Title: A Clinical Study to Evaluate the Safety and Effectiveness of the Infinity Acute Care System Workstation Neonatal Care Babylog VN500 Device in High Frequency Oscillatory Ventilation (HFOV) Mode in Very Low Birth Weight (VLBW) Neonates
Brief Title: Safety and Efficacy Study of the Draeger Babylog VN500 Device in HFOV Mode in VLBW Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Draeger Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I100738
Record Dates: First submitted 2015-05-05; First posted 2015-05-15 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Distress Syndrome In Premature Infants
Keywords: High Frequency Oscillatory Ventilation; Infant, Very Low Birth Weight; Periventricular Leukomalacia; Intraventricular Hemorrhage; multi-center study
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Leukomalacia, Periventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Babylog VN500 in HFOV mode (Experimental): Subjects will be treated with HFOV provided by the Babylog VN500 - the investigational device - for up to 14 days.
  Interventions: Device: Babylog VN500 in HFOV Mode

INTERVENTIONS:
Device: Babylog VN500 in HFOV Mode — Treatment with high frequency oscillatory ventilation with investigational device for up to 14 days

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the Babylog VN500 in high frequency oscillatory ventilation (HFOV) mode as a method for treating very low birth weight (VLBW) neonates requiring invasive respiratory support in the treatment of respiratory distress.

DETAILED DESCRIPTION:
Results from this single-arm, multi-center clinical study are intended to evaluate the safety and effectiveness of the Babylog VN500 device in high frequency oscillatory ventilation (HFOV) mode in very low birth weight (VLBW) neonates of 23 to 30 weeks' gestational age (400 g to 1200 g, inclusive) with documented respiratory distress requiring invasive respiratory support. The safety will be determined by evaluating the rate of subjects alive at Day 32 and free of Grade III/IV intraventricular hemorrhage (IVH) or cystic periventricular leukomalacia. Evaluation of the Alveolar-arterial (A-a) gradient 12 hours after start of ventilation will account for the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age between 23 to 30 weeks; within first 4 days of life
* very low birth weight between 400 g and 1200 g, inclusive
* 5-minute Apgar score >3
* documented respiratory distress requiring invasive respiratory Support
* A priori: primary intention for either HFOV or high-frequency jet ventilation OR Severity of Illness: mechanical ventilation with a fraction of inspired oxygen of ≥ 0.25% and a mean airway pressure of ≥ 7 cm H2O, more than 2 hours after an initial dose of surfactant required and clinical care team believes that treatment with HFOV is indicated
* anticipated availability of investigational device at the study center before screening for enrollment
* written informed consent to participate in the study provided by a parent or legal guardian

Exclusion Criteria:

* anticipation to require intubation and mechanical ventilation for less than 12 hours
* previous exposure to any mechanical ventilation for ≥ 96 hours before planned HFOV treatment
* obvious chromosomal or major congenital abnormalities involving the respiratory tract or upper airway
* known congenital heart disease, excluding Patent Ductus Arteriosus (PDA), ventricular-septal defect, or atrial-septal defect
* pre-existing air leak, including pneumothorax, pneumomediastinum, pneumopericardium, or extensive bilateral Pulmonary Interstitial Emphysema (PIE)
* severe metabolic acidosis with a base deficit of ≥ 15 before planned HFOV treatment
* severe hypotension (a mean blood pressure more than 2 standard deviations below the mean neonate's birth weight despite a total combined dose of dopamine, dobutamine, or both, of 20 µg(kg/min)
* moribund subject not expected to survive, or a subject in whom there is a decision to limit care
* currently receiving or previous treatment with inhaled nitric oxide
* currently receiving or previous treatment with corticosteroids specifically for BPD prevention
* evidence of severe sepsis (neutropenia, severe hypotension, shock)
* evidence of Nectrotising Enterocolitis (NEC), defined as Modified Bell's Stage II or greater
* documented Grade III/IV intraventricular hemorrhage
* current enrollment in another Investigational Device Exemption or Investigational New Drug clinical study where treatment, testing, or follow-up may interfere with the results

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Alive and free from Grade III/IV intraventricular hemorrhage (IVH) and cystic periventricular leukomalacia (PVL) | Day 32 +/- 10 days gestational age
  Papile's grading on cranial ultrasound
Alveolar-arterial (A-a) Gradient change | 12 hours after onset of HFOV treatment
  A-a Gradient as measured by arterial blood gas after onset of Treatment with the Babylog VN500 in HFOV mode

SECONDARY OUTCOMES:
Freedom from study-defined serious adverse events | during Treatment Phase (up to 14 days)
  Events related to the Condition of Prematurity and the requirement for invasive respiratory suppport
Device failure rate | during Treatment Phase (up to 14 days)
  malfunction of the investigational device necessitating removal of a neonate to another Ventilation mode or ventilator
Neurodevelopment assessment | 22 - 24 months corrected age
  Bayley Scales of Infant and Toddler Development III
Change of partial carbon dioxide pressure (PaCO2) | 2, 6, 12, 24, 36 and 48 hours after onset of HFOV treatment
  Duration of time and amount that the carbon dioxide Tension values are outside the target range of 40 to 55 mmHg
Relationship between tidal volume high frequency (Vthf) set and Vthf observed | 2, 6, 12, 24, 36 and 48 hours and once daily after onset of HFOV treatment
  difference between mean Vthf set and mean Vthf observed
Stability of Vthf observed and carbon dioxide diffusion (DCO2) coefficient monitoring during high frequency oscillation over time | first 48 hours of HFOV treatment
  this outcome will be evaluated during periods when no changes to ventilator settings are made. During the first 48 hours of treatment with the investigational device, ventilator settings, VThf and DCO2 will be downloaded from the ventilator's memory along with Ventilator settings for subsequent analysis.
Freedom from Bronchopulmonary Dysplasia (BPD) | 36 week's corrected age
  Need for any oxygen or positive airway pressure
Length and Type of Respiratory Support | participants will be followed for the duration of hospital stay, an expected average of 14 weeks
  invasive ventilator support, supplemental oxygen, positive pressure support
Neonatal survival | participants will be followed for the duration of hospital stay, an expected average of 14 weeks
  survival with and without the need for supplemental oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Martin Keszler, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (14):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - St. Paul Children's Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - North Central Baptist Hospital, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health Science Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No